CLINICAL TRIAL: NCT05372809
Title: Closure Obtained With Vascularized Epithelial Regeneration for DFUs With SkinTE®
Brief Title: Multi-Center, Prospective, Randomized Controlled Trial Evaluating SkinTE® in the Treatment of Wagner 2 DFUs
Acronym: COVER DFUs
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study terminated due to slow enrollment and change in strategy.
Sponsor: PolarityTE (Industry)
Collaborators: Alira Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: COVER DFUs
Record Dates: First submitted 2022-05-06; First posted 2022-05-13 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Diabetic Foot
Keywords: diabetic foot ulcer; regenerative medicine; SkinTE; skin regeneration; chronic wounds; Wagner 2
MeSH Terms: conditions — Diabetic Foot | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: mult-center, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the test article, a placebo harvest procedure or placebo treatment is not possible. Patients will be treated by an unblinded investigator. Wounds will be assessed at each visit by a blinded assessor. Wound closure determined by the blinded assessor will be confirmed by a blinded adjudicator.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- SkinTE (Experimental): SkinTE plus standard care
  Interventions: Biological: SkinTE
- Control (Other): Standard care alone
  Interventions: Other: Control

INTERVENTIONS:
Biological: SkinTE — SkinTE is an Autologous Heterogeneous Skin Construct (AHSC), which is manufactured from a small piece of healthy full-thickness skin harvested from the patient at the time of randomization to the SkinTE arm. SkinTE is manufactured aseptically by PolarityTE following current Good Manufacturing Practice (cGMP). SkinTE is not cultured ex vivo; rather, it is returned to the provider expeditiously to maintain cellular viability. SkinTE includes various multicellular segments as a result of the manufacturing process. The different multicellular segments contain different types of skin cells, such as keratinocytes, dermal fibroblasts, dermal endothelial cells, and follicular cells, as well as extracellular matrix. The multicellular segments have a surface area-to-volume ratio for improved sustenance by imbibition prior to engraftment.
  Other Names: Autologous Heterogeneous Skin Construct
  Arms: SkinTE
Other: Control — Standard care is defined in this protocol to include the following:
  * Debridement
  * Collagen-alginate primary wound dressing
  * Local offloading with felt pad for wounds on weight bearing surfaces
  * Foam
  * Multi-layer compression dressing
  * Off-loading device such as a full-length boot or total contact cast (if full-length boot cannot accommodate the patient) or surgical shoe for ulcers in non-weight bearing locations
  Other Names: Standard of Care
  Arms: Control

SUMMARY:
The purpose of this study is to assess the safety and efficacy of SkinTE for treatment of Wagner grade 2 diabetic foot ulcers.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized controlled trial (RCT) designed to assess the safety and efficacy of SkinTE with standard of care (SOC) dressings compared to SOC dressings alone (wound debridement, collagen-alginate dressing, multi-layer compression dressings, and offloading) in the treatment of Wagner grade 2 diabetic foot ulcers (DFUs) ranging in size from 1 to 10 cm2. After being informed about the study and potential risks, all patients giving written informed consent who meet eligibility criteria will undergo a 2-week screening period of SOC. Patients meeting eligibility criteria following the screening period will be randomized in a single-blind manner (blinded evaluator with closure confirmed by a blinded adjudicator) in a 1:1 ratio to SkinTE with SOC or SOC alone. Patients will be followed weekly for 6 months for wound closure.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Documented history of Type I or Type II Diabetes Mellitus requiring oral and/or insulin replacement therapy.
* Presence of a DFU Wagner 2 grade wound on any aspect of the foot, provided that if the malleolus is involved, not more than 50% of the wound is above the mid-point of the medial malleolus. [NOTE: DFU must maintain Wagner 2 Grade for the duration of study run-in period - i.e., screening visit 1 (SV1) to randomization visit 1 (RV1).]
* If other wounds are present on the same foot, they must be more than 2 cm distant from the index ulcer. [NOTE: If two or more DFUs are present with the same grade, the index ulcer is the largest ulcer and the only one evaluated in the study.]
* Index ulcer (i.e., current episode of ulceration) has been present for ≥ four weeks (≥ 28 days) prior to the initial screening visit (SV1).
* Index ulcer (post-debridement) is a minimum of 1.0 cm2 and a maximum of 10 cm2 at the first screening visit (SV1) and first randomization visit (RV1).
* Adequate circulation to the affected foot as documented by a dorsal transcutaneous oxygen measurement (TCOM) or a skin perfusion pressure (SPP) measurement of ≥ 30 mmHg, or an Ankle Branchial Index (ABI) of ≥ 0.7 and ≤ 1.2 or Arterial Doppler with a minimum of biphasic flow or Toe Brachial Index (TBI) ≥ 0.75 at SV1, using the affected study extremity within 30 days of screening visit (SV1).
* Index ulcer and/or index ulcer limb may have had prior infection(s), but infection(s) must be adequately treated and controlled as defined by IDSA Guidelines PEDIS Grade level 1.
* The index ulcer has been offloaded with protocol defined offloading device throughout the study run-in period for at least 14 days prior to randomization (Run- in period defined as Screening through RV1/Randomization).
* Negative pregnancy test for females of childbearing potential (e.g., not post- menopausal for at least one year or surgically sterile).
* Subject understands and is willing to participate in the clinical study and can comply with weekly visits and the follow-up regimen.
* Females of childbearing potential must agree to use effective methods of contraception (birth control pills, barriers, or abstinence) (Screening through End of Study (EOS) and undergo pregnancy tests.
* Properly obtained written informed consent.
* Subject must have stable living environment in order to manage offloading and wound care management.
* The index ulcer has a clean base, free of necrotic debris, and infection at time of placement of treatment product.

Exclusion Criteria:

* Index ulcer and/or index limb with presence of gangrene or unstable ischemia at screening (SV1).
* Revascularization surgery on the lower extremity on which the index ulcer is located within 30 days of screening (SV1).
* Index ulcer in the opinion of the investigator, is suspicious for cancer and should undergo an ulcer biopsy to rule out a neoplasm of the ulcer.
* Subjects with history of radiation on the same limb as the index ulcer (regardless of time since last radiation treatment).
* Subjects with exposed internal fixation on the same limb as the index ulcer. [NOTE: External fixation is allowed if deemed stable by principal investigator.]
* Subjects on any investigational drug(s) or therapeutic device(s) within 30 days preceding the first screening visit (SV1). ). [NOTE: NPWT is allowed up to the day of screening (SV1), if in the opinion of the Principal Investigator NPWT may be discontinued.]
* Index ulcer treated within the last 30 days prior to screening with a prohibited treatment as defined in full protocol.
* Subjects with a history of more than two weeks treatment with immunosuppressants (including systemic corticosteroids > 10mg prednisone (or equivalent) daily dose), cytotoxic chemotherapy, or application of topical steroids to the index ulcer surface within 30 days prior to first screening visit (SV1), or who receive such medications during the run-in period, or who are anticipated to require such medications during the study.
* Presence of any condition(s) which seriously compromises the subject's ability to complete this study or has a known history of poor adherence to medical treatment.
* In the opinion of the investigator, the subject is non-compliant with offloading or index ulcer dressing during the run-in period.
* Active Charcot's arthropathy of the index ulcer limb as verified by clinical evaluation, and/or imaging (x-ray or MRI) within 30 days prior to randomization (RV1).
* Subjects with chronic osteomyelitis and/or cellulitis on the same limb as the index ulcer as verified by clinical evaluation, and/or imaging (x-ray or MRI) within 30 days prior to randomization (RV1).
* Subject is pregnant or breast-feeding.
* Presence of diabetes with poor metabolic control as documented as not having at least one HbA1c ≥12.0 within 30 days prior to randomization (RV1).
* Subjects with end stage renal disease requiring treatment with dialysis and/or evident by an eGFR <30 mL/min/1.73m2 within 120 days of randomization (RV1). [NOTE: Subjects with two documented eGFR values within 120 days, the most recent value may be used if the eGFR ≥30 mL/min/1.73m2 and is, in the opinion of the principal investigator, stable and the subject will not require treatment with dialysis for the duration of study participation.]
* Index ulcer has reduced or increased in area by 30% or more after 14 days of SOC from SV1 to the RV1/randomization visit.
* Evidence of unstable human immunodeficiency virus (HIV), hepatitis B, and/or hepatitis C in the opinion of the investigator at first screening visit (SV1).
* Documented history of New York Heart Association Class III or IV congestive heart failure or unstable cardiovascular disease requiring intervention within 60 days prior to screening (SV1).
* Requiring surgical intervention (excluding debridement) at the time of consenting and/or increased probability of requiring surgical intervention during study participation [NOTE: non-invasive surgical intervention is allowed if, per the Principal Investigator, treatment will not affect subject's ability to participate in clinical trial.]
* Any clinically significant finding, in the judgment of the investigator, that would place the subject at health risk, impact the study, or affect the completion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-02-21 (Actual); Study Completion 2024-02-21 (Actual)

PRIMARY OUTCOMES:
Incidence of index ulcers closed | 24 weeks
  Wound closure is confirmed at two consecutive visits each two weeks apart

SECONDARY OUTCOMES:
Percent area reduction (PAR) | Assessed at 4, 8, 12, 16, 20, and 24 weeks
  Change in wound area from the time of randomization
Incidence of index ulcers closed | 12 weeks
  Wound closure is confirmed at two consecutive visits each two weeks apart
Time to closure | up to 24 weeks
Wound Quality of Life (w-QoL) Questionnaire | 24 weeks
  Change in w-QoL from baseline
Wound infection | 24 weeks
  Incidence of new onset infection of index ulcer requiring treatment with antibiotics

OTHER OUTCOMES:
Incidence of pain, infection, and complications of the harvest site | 24 weeks
Incidence of adverse events of the index ulcer | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nikolai Sopko, MD, PhD, Study Director — PolarityTE; David Armstrong, DPM, MD, PhD, Study Chair — University of Southern California; Lawrence Lavery, DPM, Principal Investigator — University of Texas
Locations (13):
- United States (13):
  - Limb Preservation Platform, INC, Fresno, California
  - LA Foot and Ankle Clinic, Los Angeles, California
  - Royal Research, Corp, Hollywood, Florida
  - Barry University Clinical Research, Tamarac, Florida
  - Gateway Clinical Trials, O'Fallon, Illinois
  - Boston Medical Center, Boston, Massachusetts
  - Mount Sinai West, New York, New York
  - Northwell Health, New York, New York
  - VA North Texas Health Care System, Dallas, Texas
  - University of Texas Southwestern Wound Care Clinic, Dallas, Texas
  - Futuro Clinical Trials, LLC, McAllen, Texas
  - Baylor Scott & White Research Institute - Plano, Plano, Texas
  - Foot and Ankle Institute, St. George, Utah